CLINICAL TRIAL: NCT01137318
Title: Combined Cognitive Remediation and Behavioral Intervention for Treatment of ADHD
Brief Title: Combined Cognitive Remediation and Behavioral Intervention for Treatment of Attention-deficit/Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queens College, The City University of New York (Other)
Responsible Party: Principal Investigator, Anil Chacko, Assistant Professor, Queens College, The City University of New York
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R34MH088845-01 (NIH)
Record Dates: First submitted 2010-02-24; First posted 2010-06-04 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: ADHD
Keywords: ADHD; Impairment; Treatment; Cognitive Remediation; Behavioral Parent Training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive remediation and Behavioral Intervention (Experimental)
  Interventions: Behavioral: Cognitive remediation and Parent Training
- Low Level Cognitive Remediation and Behavioral Parent Traning (Placebo Comparator)
  Interventions: Behavioral: Cognitive remediation and Parent Training

INTERVENTIONS:
Behavioral: Cognitive remediation and Parent Training — Cognitive Intervention is CogMed Working Memory Training program, which is a 5-week, 5days/week computerized training program completed at home. The Parent Training is a 2.0 hour, weekly, group sessions that focus on behavioral management procedures.

SUMMARY:
The objective of this study is to evaluate a novel sequenced combination of a promising, computerized cognitive training program targeting working memory (WM) deficits in children with attention-deficit/hyperactivity disorder (ADHD) in combination with behavioral parent training, a well-established, evidence-based intervention for ADHD.

The combined active intervention, compared to the combined control intervention will result in improvement in primary psychosocial (i.e., parent/teacher reported child impairment; parental stress; parenting behavior; and observed child academic achievement) and psychiatric (parent/teacher rated ADHD, ODD, and CD symptoms; observed activity level and attention) outcomes at post-treatment and follow up assessment, with the combined active intervention resulting in greater improvements in these outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of ADHD Children 7-11 year olds English Speaking

Exclusion Criteria:

- Pervasive Developmental Disorder IQ< 80

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
ADHD Symptoms | 3 month follow up
  Disruptive Behavior Disorder Rating Scale: ADHD symptoms will be measured using the Disruptive Behavior Disorders rating scale (DBD) administered to the child's parent and teacher. The DBD is a 45-item measure that asks parents to rate the DSM symptoms of ADHD, ODD, and CD on a four point Likert scale (i.e., Not at all, Just a little, Pretty Much, or Very Much). For this study, the average scores for DSM-IV Inattentive symptoms, DSM-IV Hyperactive-Impulsive symptoms, DSM-IV ODD symptoms, and DSM-IV CD symptoms will be used.
Impairment | 3 month follow up
  Parent and teacher ratings of problem severity and need for treatment in important functional domains will be measured using the Impairment Rating Scale (IRS). The IRS measures impairment across domains of functioning as well as overall need for treatment. Parents and teachers place an "x" on a seven-point visual analogue scale to signify their child's functioning along a continuum of impairment that ranges from zero (Not a problem at all. Definitely does not need treatment or special services.) to six (Extreme problem. Definitely needs treatment and special services).
Academic Achievement | 3 month follow up
  Wide Range Achievement Test 4 Progress Monitoring Version [WRAT4-PMV]is an adaptation of the WRAT4 and is specifically designed to be a reliable and efficient tool for monitoring the academic progress of students in Grades K-12 and college. A series of brief 15-item tests are offered in 4 areas of basic skills: word reading, sentence comprehension, spelling, and mathematics computation.
ODD symptoms | 3 month follow up
  Disruptive Behavior Disorder Rating Scale: ODD symptoms will be measured using the Disruptive Behavior Disorders rating scale (DBD) administered to the child's parent and teacher. The DBD is a 45-item measure that asks parents to rate the DSM symptoms of ADHD, ODD, and CD on a four point Likert scale (i.e., Not at all, Just a little, Pretty Much, or Very Much). For this study, the average scores for DSM-IV Inattentive symptoms, DSM-IV Hyperactive-Impulsive symptoms, DSM-IV ODD symptoms, and DSM-IV CD symptoms will be used.
CD symptoms | 3 month follow up
  Disruptive Behavior Disorder Rating Scale:CD symptoms will be measured using the Disruptive Behavior Disorders rating scale (DBD) administered to the child's parent and teacher. The DBD is a 45-item measure that asks parents to rate the DSM symptoms of ADHD, ODD, and CD on a four point Likert scale (i.e., Not at all, Just a little, Pretty Much, or Very Much). For this study, the average scores for DSM-IV Inattentive symptoms, DSM-IV Hyperactive-Impulsive symptoms, DSM-IV ODD symptoms, and DSM-IV CD symptoms will be used.
Motor Activity | 3 month follow up
  Solid-state actigraph: Motor activity will be recorded throughout the assessment using two solid-state actigraphs that store data on the number of movements per unit time. Actigraphs will be worn on the waist and non-dominant ankle. Assessments of activity level taken during structured test-sessions in children are reliable and yield measures that are correlated with parent and teacher ratings of hyperactivity
Inattention | 3 month follow up
  A-X Continuous Performance Test CPT214: This CPT runs on a computer and generates objective measures of inattention and impulsivity. Letters are presented individually for 200 msec., with a 1.5 sec. interstimulus interval. The child responds when he sees an "A" followed by an "X". A total of 400 letters are presented and the entire task lasts approximately 12 minutes.
Impulsivity | 3 month follow up
  A-X Continuous Performance Test CPT214: This CPT runs on a computer and generates objective measures of inattention and impulsivity. Letters are presented individually for 200 msec., with a 1.5 sec. interstimulus interval. The child responds when he sees an "A" followed by an "X". A total of 400 letters are presented and the entire task lasts approximately 12 minutes.
Parenting Behavior | 3 month follow up
  Alabama Parenting Questionnaire: The Alabama Parenting Questionnaire (APQ) is a 42-item measure of parenting that asks parents to rate different domains of parenting on a five-point scale ranging from one (never) to five (always). The APQ can be divided into six scales: Involvement, Positive Parenting, Poor Monitoring/Supervision, Inconsistent Discipline, Corporal Punishment, and an Other Discipline Practices Scale.
Parenting Stress | 3 month follow up
  Parenting Stress Index-Short Form (PSI-SF). To gather information concerning the degree of and types of stress attributed to parenting, each parent will complete the PSI-SF. The PSI-SF is a direct derivative of the full-length test and consists of a 36-item self-scoring questionnaire/profile. It yields a Total Stress score from 3 scales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child

CONTACTS AND LOCATIONS:
Overall Officials: Anil Chacko, PhD, Principal Investigator — Queens College, The City University of New York
Locations (1):
- Queens College, Flushing, New York, United States

REFERENCES:
- [Derived] Chacko A, Bedard AC, Marks DJ, Feirsen N, Uderman JZ, Chimiklis A, Rajwan E, Cornwell M, Anderson L, Zwilling A, Ramon M. A randomized clinical trial of Cogmed Working Memory Training in school-age children with ADHD: a replication in a diverse sample using a control condition. J Child Psychol Psychiatry. 2014 Mar;55(3):247-55. doi: 10.1111/jcpp.12146. Epub 2013 Oct 7. PMID 24117656
- See also: Refining Attention Memory and Parenting Study for Youth with ADHD — http://www.chipslab.org/news/RAMP/